CLINICAL TRIAL: NCT05023343
Title: Does Administration of the Transmuscular Quadratus Lumborum Block Cause Quadriceps Muscle Weakness: A Randomised, Double-blinded Volunteer Study
Brief Title: Transmucular Quadratus Lumborum Block: Potential Quadriceps Muscle Weakness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUH-TQL-QUADRICEPS
Record Dates: First submitted 2021-08-17; First posted 2021-08-26 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Neuromuscular Blockade
Keywords: Quadratus lumborum; Quadratus lumborum block; Ultrasound; Muscle weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Ropivacaine; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Each participant serves as their own control i.e. each participant will receive both an active and placebo block TQL block. Left/right side are randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Unilateral transmuscular quadratus lumborum block using 30 mL 0.75% ropivacaine
  Interventions: Drug: Ropivacaine; Other: Quadriceps muscle strength; Other: Timed Up and Go; Other: Single-leg 6 meter timed hop test; Other: Temperature discrimination; Other: Pinprick test; Diagnostic Test: Blood samples; Diagnostic Test: Non-invasive blood pressure measurement
- Placebo (Placebo Comparator): Unilateral transmuscular quadratus lumborum block using 30 mL isotonic saline
  Interventions: Other: Quadriceps muscle strength; Other: Timed Up and Go; Other: Single-leg 6 meter timed hop test; Other: Temperature discrimination; Other: Pinprick test; Diagnostic Test: Blood samples; Diagnostic Test: Non-invasive blood pressure measurement

INTERVENTIONS:
Drug: Ropivacaine — 30 mL Ropivacaine 0,75% administered as a unilateral TQL block
  Arms: Active
Other: Quadriceps muscle strength — Quadriceps muscle strength is assessed using a hand-held dynamometer. Each participant is tested pre block administration and 60 minutes after
Other: Timed Up and Go — To test mobilisation the standardised Timed Up and Go test is used. Each participant is tested pre block administration and 60 minutes after
Other: Single-leg 6 meter timed hop test — To test muscle strength and power the single-leg 6 meter jump test is used. Each participant is tested pre block administration and 60 minutes after
Other: Temperature discrimination — Dermatomal evaluation of cold and warm discrimination of the thoracic and lumbar dermatomes Approximately 60 minutes after block administration
Other: Pinprick test — Dermatomal evaluation of pinprick/sharp sensation of the thoracic and lumbar dermatomes.
  Approximately 60 minutes after block administration
Diagnostic Test: Blood samples — As a substudy the maximum serum concentration of ropivacaine is analyzed. Blood samples are taken at 0, 15, 30, 45 and 60 minutes after block administration
Diagnostic Test: Non-invasive blood pressure measurement — Non-invasive blood pressure is measured prior to block administration and 30 minutes after block administration

SUMMARY:
The aim of this study is to examine whether the administration of the TQL block cause motor block of the lumbar plexus and thereby quadriceps muscle weakness. The investigators hypothesise that the administration of a unilateral TQL block does not cause quadriceps muscle weakness compared to a placebo block.

DETAILED DESCRIPTION:
The ideal postoperative analgesic regimen following major abdominal and retroperitoneal laparoscopic surgery still lacks consensus and the discussion is ongoing. The epidural blockade has been the gold standard for postoperative pain management for major abdominal surgery for years, but with the conversion to minimal invasive surgery the procedure can rarely be justified.

The use of a multimodal analgesic regimen with opioids can cause severe side effects. These side effects can delay mobilisation after surgery, increase the risk of complications and worst of all be fatal.

The focus on an opioid sparing regimen, in the enhanced recovery setting, has been a significant motivator for the addition of ultrasound-guided nerve blocks to the perioperative progression.

At the Department of Anaesthesiology, Zealand University Hospital, the ultrasound-guided Transmuscular Quadratus Lumborum (TQL) block is part of the perioperative pain regimen for major laparoscopic abdominal and retroperitoneal surgeries, as well as for elective caesarean sections. Using the visual guidance of ultrasound, the injectate of local anaesthetic is administered in the fascial interspace between the quadratus lumborum muscle and the psoas major muscle posterior to the transversalis fascia.

This will anaesthetise the abdominal wall including both somatic and visceral nerves. No involvement of lumbar plexus i.e. the femoral nerve, obturator nerve or the lumbar part of the sympathetic trunk was observed. The lack of lumbar plexus involvement means no motor block of the lower extremities should be observed. Previous clinical studies reported no adverse events. However, the investigators did not specifically register lower limb weakness or hypotension, but on the other hand did not find any difference in ambulation or even faster ambulation compared to the placebo group.

A few case reports have reported complications related to the various quadratus lumborum blocks. Ueshima et al. reported that 90% (65/81 cases) experienced quadriceps muscle weakness following a TQL block. The incidence was 19% for posterior QL block and 1% for lateral QL block. Lower limb weakness was also reported by Wikner et al. following a bilateral lateral QL block. A case of continuous hypotension after administration of a lateral QL block has been described. One case of unilateral upper limb weakness and Horners Syndrome after a bilateral posterior QL block has also been reported. Urinary retention was reported following a continuous TQL-block. All side effects were temporary, no one reported permanent injuries. Complications have not been reported systematically.

At Zealand University Hospital, Roskilde, the investigators have administrated more than 1000 TQL blocks, and more than 300 patients have been included in various clinical trials. From clinical experience and cadaveric studies, the investigators find no evidence that the TQL block spread to the epidural space, and therefore does not cause sympathetic symptoms. Neither does the TQL block spread to the lumbar plexus, and therefore does not cause motor weakness of the lower extremities. However these notions have never been properly investigated in a controlled clinical setting, meaning that the investigators cannot entirely rule out the possibility of a spread to the lumbar plexus and thus ensuing quadriceps muscle weakness. This calls for a more in-depth investigation of this potential phenomenon.

Therefore, the aim of this study is to examine whether the administration of the TQL block cause motor block of the lumbar plexus and thereby quadriceps muscle weakness.

Prior to block administration all participants are tested using the same motor tests as after the block administration(baseline tests).

All participants will receive two TQL blocks. To keep participants and outcome assessors blinded the study drug for each side will be randomised i.e. active treatment on one side and placebo on the contralateral side.

The investigators hypothesise that the administration of a unilateral TQL block does not cause quadriceps muscle weakness compared to a placebo block.

Sub-study:

Fascial plane nerve blocks demand a great volume of local anaesthetic to achieve the right spread of local anaesthetic and thus a sufficient analgesia.

The correct concentration and volume of local anaesthetic is still debated. Studies measuring serum concentrations of local anaesthetic are rare due to time consumption and high costs. When administering a unilateral TQL block a volume of 30 ml local anaesthetic is used often equal to the maximum single-shot dose of ropivacaine; i.e. 225 milligrams. In previous studies and in the usual clinical setting the investigators have never experienced any signs of systemic toxicity, however the maximum serum concentration of local anaesthetic following TQL block administration has never been investigated. The maximum serum ropivacaine concentration following administration of a TQL block will therefore be investigated for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* American Associations of Anaesthesiologist (ASA) class 1-2
* Have received written and oral information and signed the consent form
* Weight > 56,5 kilograms (Chosen due to maximum single dose of ropivacaine i.e. 225 milligrams)

Exclusion Criteria:

* Inability to speak and understand Danish
* Inability to cooperate
* Allergy to study drugs
* Daily intake of opioids
* Alcohol and/or drug overuse
* Fertile female participants: No use of safe contraceptives for the last month, positive urine-HCG or breastfeeding
* Previous trauma of surgery in the abdomen, hip or knee.
* Any systemic muscular or neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Maximum unilateral knee extension strength | One hour
  The change in maximum, unilateral knee extension strength (newtonmeters (Nm)) comparing active and placebo TQL block, measured as the change from baseline to one hour after block administration.

SECONDARY OUTCOMES:
Single-leg 6 meter timed hop test | One hour
  Change in time performing the single-leg 6 meter timed hop test (Minutes, standardised protocol) comparing active and placebo TQL block, measured as the change from baseline to one hour after block administration.
Timed Up and Go test | One hour
  Change in Timed Up and Go test (minutes, standardised protocol) from baseline to one hour after block administration
Dermatomal testing of thoracic and lumbar dermatomes | One hour
  Dermatomal spread of the TQL block using standardised mechanical (pinprick) discrimination (number of dermatomes)
Dermatomal testing of thoracic and lumbar dermatomes | One hour
  Dermatomal spread of the TQL block using standardised temperature (cold) discrimination (number of dermatomes).
Dermatomal testing of thoracic and lumbar dermatomes | One hour
  Dermatomal spread of the TQL block using standardised temperature (warmth/heat) discrimination (number of dermatomes).
Non-invasive blood pressure (Mean arterial pressure) | 30 minutes
  Change in non-invasive blood mean arterial pressure from baseline to T30min (mmH
Adverse events | At least 2 hours post block administration
  Number of adverse events
Total ropivacaine serum concentration | One hour
  Total concentration of ropivacaine at 0, 15, 30, 45 and 60 minutes following administration of the unilateral TQL block.

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Tanggaard, MD, Principal Investigator — Zealand University Hospital, Department of Anaesthesiology
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, Zealand University Hospital, Roskilde, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanggaard K, Nielsen MV, Holm UHU, Hoffmann BM, Bernhoff C, Andersen CH, Thomassen SS, Hansen C, Dam M, Poulsen TD, Holm PM, Borglum J. No quadriceps muscle weakness following anterior quadratus lumborum block compared with placebo: a randomized, non-inferiority, blinded, volunteer trial. Reg Anesth Pain Med. 2025 Jul 4;50(7):568-574. doi: 10.1136/rapm-2024-105313. PMID 38754991